CLINICAL TRIAL: NCT01462812
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Evaluating the Efficacy and Safety of a Single 20 mg Dose of Sumatriptan Powder Delivered Intranasally With the Bi-directional Device in Adults With Acute Migraine With or Without Aura
Brief Title: Safety & Efficacy of a Single Dose of Sumatriptan Powder Delivered Intranasally With the Bi-directional Device in Adults With Acute Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Optinose US Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPN-SUM-MIG-3301
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Results first posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2012-08

CONDITIONS: Migraine Headache
Keywords: Migraine; Headache; Sumatriptan
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sumatriptan (Active Comparator)
  Interventions: Drug: Sumatriptan
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sumatriptan — Sumatriptan 20mg
  Arms: Sumatriptan
Drug: Placebo — Matching placebo
  Arms: Matching placebo

SUMMARY:
The study is being conducted to determine if OPTINOSE SUMATRIPTAN delivered nasally (through the nose) using the OPTINOSE SUMATRIPTAN Device can reduce the pain and symptoms associated with migraine headaches.

DETAILED DESCRIPTION:
The primary objective for this study is to compare headache relief (defined as a reduction from moderate [Grade 2] or severe [Grade 3] pain to none [Grade 0] or mild [Grade 1] pain) at 120 minutes following a dose of 20 mg of OPTINOSE SUMATRIPTAN with placebo in the acute treatment of a single migraine attack.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, between the ages of 18 to 65 years
* Diagnosis of migraine, with or without aura
* Experiences between 1 and 8 migraine attacks per month for the past 12 months

Exclusion Criteria:

* Inability to distinguish other headaches from migraine
* Experiences headache of any kind at a frequency greater than or equal to 15 days per month
* History of resistance to sumatriptan, or non-response to 2 or more other triptans, defined as subjects who have not responded to an adequate dose and duration of treatment
* Current use of medication for migraine prophylaxis that has not been stable (no dose adjustment) for 30 days prior to screening
* Chronic opioid therapy (>3 consecutive days in the 30 days prior to screening)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - San Francisco Clinical Research Center, San Francisco, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Associated Neurologists of Southern CT, P.C., Fairfied, Connecticut
  - Premiere Research Institute, West Palm Beach, Florida
  - MedVadis, Watertown, Massachusetts
  - Michigan Head and Pain Institute, Ann Arbor, Michigan
  - ClinVest, Springfield, Missouri
  - Mercy Health Research, St Louis, Missouri
  - DENT Neurologic Institute, Amherst, New York
  - Headache Wellnes Center, Greensboro, North Carolina
  - PMG Research of Raleigh North carolina, LLC, Raleigh, North Carolina
  - PMG Research of Winston Salem, LLC, Winston-Salem, North Carolina
  - Neurology Center of Ohio, Toledo, Ohio
  - Jefferson Headache Center, Philadelphia, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina

REFERENCES:
- [Derived] Cady RK, McAllister PJ, Spierings EL, Messina J, Carothers J, Djupesland PG, Mahmoud RA. A randomized, double-blind, placebo-controlled study of breath powered nasal delivery of sumatriptan powder (AVP-825) in the treatment of acute migraine (The TARGET Study). Headache. 2015 Jan;55(1):88-100. doi: 10.1111/head.12472. Epub 2014 Oct 30. PMID 25355310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: private practices and research clinics
Pre-assignment Details: Screening period (general medical exams, labs, medical and headache history, concomitant medications.
Groups:
- Matching Placebo: Placebo : Matching placebo
- Sumatriptan: Sumatriptan : Sumatriptan 20mg
Period: Overall Study
Arm/Group | Matching Placebo | Sumatriptan
Started | 111 | 112
Completed | 111 | 111
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Matching Placebo | Sumatriptan | Total
Number analyzed (Participants) | 111 | 112 | 223
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 111 | 112 | 223
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (10.71) | 42.2 (10.27) | 42.2 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 94 | 187
  Male | 18 | 18 | 36
Region of Enrollment [Number; unit: participants]
  United States | 111 | 112 | 223

OUTCOME MEASURES:

1. Primary Outcome: Headache Relief
Description: The primary objective for this study is to compare headache relief (defined as a reduction from moderate [Grade 2] or severe [Grade 3] pain to none [Grade 0] or mild [Grade 1] pain) at 120 minutes following a dose of 20 mg of OPTINOSE SUMATRIPTAN with placebo in the acute treatment of a single migraine attack.
Time Frame: 120 Minutes
Population: The full analysis dataset (FAD) will include all subjects who are randomized, receive study medication, and record at least one post-treatment assessment of pain severity. The treatment group assignment will be designated according to treatment received. The FAD will serve as the basis for the efficacy analyses.
Measure: Number; unit: participants
Arm/Group | Matching Placebo | Sumatriptan
Number analyzed (Participants) | 104 | 108
participants | 47 | 73

ADVERSE EVENTS:
Time Frame: 17 months
Arm/Group | Matching Placebo | Sumatriptan
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/112
Other Adverse Events (participants affected / at risk) | 9/111 | 45/112
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Matching Placebo (N=111) | Sumatriptan (N=112)
Product Taste Abnormal (General disorders) | 4 | 25
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 2 | 15
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Rhinitis (Infections and infestations) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Found in PI contract.